CLINICAL TRIAL: NCT04882280
Title: Dose-dependent Impact of Daytime Lighting on Evening Responses to Light
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Palo Alto Veterans Institute for Research (Other)
Responsible Party: Principal Investigator, Jamie M. Zeitzer, Ph.D., Associate Professor, VA Palo Alto Health Care System
Organization: VA Palo Alto Health Care System (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Reverse DRC
Record Dates: First submitted 2021-05-07; First posted 2021-05-11 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Sleep
MeSH Terms: interventions — Light

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low room (Experimental): Low intensity (80 lux) room light
  Interventions: Behavioral: Light
- Normal room (Experimental): Normal intensity (150 lux) room light
  Interventions: Behavioral: Light
- Bright room (Experimental): High intensity (500 lux) room light
  Interventions: Behavioral: Light
- Bright (Experimental): Very high intensity (1000 lux) room light
  Interventions: Behavioral: Light

INTERVENTIONS:
Behavioral: Light — 10 hours of light exposure during the daytime, starting 2 hours after habitual wake time

SUMMARY:
The purpose of this study is to systematically examine the impact of different intensities of daytime light and the subsequent impact that such exposure has on non-image forming responses to light in the evening.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65
2. Good health
3. Male or female
4. Normal color vision

Exclusion Criteria:

1. Sleep disorders
2. Extreme chronotypes
3. Routine smoker
4. Significant hearing loss
5. Depressed
6. Alcohol use disorder
7. Use of illegal drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Suppression of melatonin production | 4 hours
  Difference in salivary melatonin concentrations between active arm and 3 lux control condition
Phase shift in the timing of melatonin onset | 2 days
  Change in the onset of melatonin secretion after experimental stimulus

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No